CLINICAL TRIAL: NCT06748040
Title: Genetic Testing to Understand and Address Renal Disease Disparities Across the United States - Pharmacogenetic Substudy
Brief Title: Genetic Testing to Understand and Address Renal Disease Disparities Across the United States Pharmacogenetic Substudy
Acronym: GUARDD-US PGx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); Icahn School of Medicine at Mount Sinai (Other); University of Florida (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102997_A; U01HG010225 (NIH); U01HG007269 (NIH); U01HG010248 (NIH); U01HG010245 (NIH)
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: Kidney Disease; Genetic testing; Pharmacogenomics; Hypertensive medications
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Immediate versus delayed return of pharmacogenetics (PGx) testing results to provider and participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Return of Results (Active Comparator): Immediate return of pharmacogenetic (PGx) results to substudy (APOL1 negative) participant.
  Interventions: Other: Timing of return of results
- Delayed Return of Results (Active Comparator): Delayed return of pharmacogenetic (PGx) results to substudy (APOL1 negative) participant until after the completion of the 6 month final study visit.
  Interventions: Other: Timing of return of results

INTERVENTIONS:
Other: Timing of return of results — Participants will be randomized to immediate versus delayed return of PGx results.

SUMMARY:
This is a substudy of GUARDD-US (Genetic testing to Understand and Address Renal Disease Disparities across the United States, NCT04191824). Its primary purpose is to determine the effect of knowledge of genetic test results that predict efficacy of various antihypertensive medications on change in SBP (systolic blood pressure) from baseline to 3 months in APOL1 (apolipoprotein L1) negative individuals at participating sites.

DETAILED DESCRIPTION:
GUARDD-US includes a substudy that randomizes participants in the Intervention arm who are from the PGx substudy participating sites and who test negative for APOL1 to PGx Intervention (i.e., immediate PGx ROR) and PGx Control (i.e., delayed PGx ROR) in a 1:1 ratio. This substudy will compare outcomes between participants in the PGx Control group and the PGx Intervention group.

New data show that genetic differences may cause patients to respond differently antihypertensive medication therapy. Pharmacogenomics may help guide initial or add-on antihypertensive therapy management. However, the impact of PGx testing on BP has not been studied in clinical trials among general or African ancestry populations.

Population for PGx Substudy:

Participants from Randomized Population who are randomized to Intervention and who test negative for APOL1. Only participants from PGx-substudy participating sites are included in this population.

Substudy Analyses:

Major primary endpoint analyses conducted for the APOL1 main study will be repeated for the PGx substudy focusing on differences in outcomes between APOL1 negative individuals with immediate PGx ROR (PGx Intervention) and APOL1 negative individuals with delayed PGx ROR (PGx Control).

ELIGIBILITY:
Inclusion Criteria:

* Self reported African ancestry
* English Speaking
* Age 18-70 years
* Have diagnosis of hypertension: Diagnosis of hypertension is defined by either:

  * ICD10 diagnosis codes (i.e., I10; I11.x; I12.x; I13.x; I16.x) OR
  * On active antihypertensive therapy for indication of hypertension OR
  * Having systolic blood pressure of 140 mm Hg or greater in at least 2 of the last 3 consecutive recorded values in the EHR OR
  * Having hypertension in the patient's medical record problem list
* Have been seen at ≥1 time in past year at a participating primary care site
* Either: 1) do not have diabetes and do not have CKD, or 2) have CKD; Participants with diabetes may be included as long as they also have CKD.

CKD is defined by either: A) ICD10 codes (i.e., N18.x; E08.22; E09.22; E10.22; E11.22;E13.22 (exclude Z94.0; N18.6; Z99.2)) OR B) Microalbumin/proteinuria level >30 mg/g for 2 time periods ≥ 3 months. Values taken within 12 months of enrollment, unless 2 values are unavailable, then review within 24 months of enrollment. OR C) 15 ≤ eGFR ≤ 60 ml/min for 2 time periods ≥ 3 months. GFRs are taken within 12 months of enrollment, unless 2 values are unavailable, then review within 24 months.

Diabetes is defined by: HbA1c ≥ 6.5 at least one time in the last year OR ICD10 diagnosis codes OR Having diabetes in the patient's medical record problem list.

Exclusion Criteria:

* Have diabetes, but no CKD.
* Are currently on dialysis (ICD 10 codes N18.6, Z99.2 and Z94.0)
* Have ESRD (eGFR<15 ml/min)
* Have a left ventricular assist device (LVAD)
* Have a terminal illness
* Have patient-reported known pregnancy at time of enrollment
* Have had a liver, kidney, or allogeneic bone marrow transplant
* Too cognitively impaired to provide informed consent and/or complete the study protocol
* Institutionalized or too ill to participate (i.e. incarcerated, psychiatric or nursing home facility)
* Plan to move out of the area within 6 months of enrollment
* Not a current patient seeing a provider who cares for their hypertension (i.e., family medicine, internal medicine, nephrology, HIV provider, cardiology, hypertension specialists) at a participating site
* Previously participated in the GUARDD pilot study OR have previously undergone APOL1 testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1874 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hrishikesh Chakraborty, DrPH, Study Director — Duke University; Carol Horowitz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida - Gainesville, Gainesville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Institute for Family Health, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Data Coordinating Center (DCC) will submit de-identified participant level datasets and associated documentation to the NHGRI's data repository - Genomic Analysis, Visualization and Informatics Lab-space (AnVIL), for use by other investigators. The datasets and associated documentation will be available after publication of the primary results manuscript. Documentation will include annotated case report forms, list of derived variables along with descriptions, and a description of the data model and de-identification process. The substudy data will be submitted within the main study complete dataset.
Supporting Information: Study Protocol, ICF
Time Frame: 3 months after publication
Access Criteria: Datasets will be designated as controlled access and researchers will be able to apply to NIH data access committees (DACs) for use of these datasets.

REFERENCES:
- [Background] Eadon MT, Cavanaugh KL, Orlando LA, Christian D, Chakraborty H, Steen-Burrell KA, Merrill P, Seo J, Hauser D, Singh R, Beasley CM, Fuloria J, Kitzman H, Parker AS, Ramos M, Ong HH, Elwood EN, Lynch SE, Clermont S, Cicali EJ, Starostik P, Pratt VM, Nguyen KA, Rosenman MB, Calman NS, Robinson M, Nadkarni GN, Madden EB, Kucher N, Volpi S, Dexter PR, Skaar TC, Johnson JA, Cooper-DeHoff RM, Horowitz CR; GUARDD-US Investigators. Design and rationale of GUARDD-US: A pragmatic, randomized trial of genetic testing for APOL1 and pharmacogenomic predictors of antihypertensive efficacy in patients with hypertension. Contemp Clin Trials. 2022 Aug;119:106813. doi: 10.1016/j.cct.2022.106813. Epub 2022 Jun 1. PMID 35660539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by providers who care for participants with hypertension (including, for example, general internists, primary care providers, and nephrologists).
Pre-assignment Details: Among the 6754 participants randomized into the GUARDD-US main trial, 1874 participants were further randomized into the GUARDD-US PGx substudy. These participants were assigned to the 'Immediate Return of Results' treatment group in the main trial, were from PGx-substudy participating sites and had an APOL1 negative phenotype. For this study, APOL1 negative refers to participants without 2 high risk alleles at the APOL1 locus also termed as without APOL1-HR.
Period: Overall Study
Arm/Group | Immediate Return of Results | Delayed Return of Results
Started | 953 | 921
Completed | 813 | 780
Not Completed | 140 | 141
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 134 | 132
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Immediate Return of Results: Immediate return of pharmacogenetic (PGx) results to substudy (APOL1 negative/without APOL1-HR) participant.
- Delayed Return of Results: Delayed return of pharmacogenetic (PGx) results to substudy (APOL1 negative/without APOL1-HR) participant until after the completion of the 6 month final study visit.
- Total: Total of all reporting groups
Arm/Group | Immediate Return of Results | Delayed Return of Results | Total
Number analyzed (Participants) | 953 | 921 | 1874
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (10.4) | 54.7 (11.0) | 55.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 610 | 590 | 1200
  Male | 343 | 331 | 674
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 35 | 67
  Not Hispanic or Latino | 917 | 879 | 1796
  Unknown or Not Reported | 4 | 7 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 0 | 2
  Race: Asian | 1 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Race: Black or African American | 852 | 828 | 1680
  Race: White | 0 | 0 | 0
  Race: North African/Mediterranean | 0 | 1 | 1
  Race: More than one race | 65 | 60 | 125
  Race: Unknown or Not Reported | 31 | 32 | 63
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 953 | 921 | 1874

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Baseline to 3 Months for APOL1 Negative Participants
Time Frame: Baseline to 3 month study visit
Population: Intent To Treat (ITT) population for PGx substudy.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Return of Results | Delayed Return of Results
Number analyzed (Participants) | 877 | 830
mmHg | -3.7 (19.0) | -3.1 (19.0)
Statistical Analysis 1: Comparison: Immediate Return of Results vs Delayed Return of Results; Test type: Superiority; p = 0.4852, t-test, 2 sided — P-value less than 0.05 is considered as statistically significant; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.4 to 1.2]

ADVERSE EVENTS:
Time Frame: 6 months
Description: GUARDD-US does not include a drug or device intervention. For this reason, no adverse events (other than all-cause mortality) were collected or recorded in the study database.
Arm/Group | Immediate Return of Results | Delayed Return of Results
All-Cause Mortality (participants affected / at risk) | 3/953 | 4/921
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT06748040/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT06748040/ICF_001.pdf